CLINICAL TRIAL: NCT00740519
Title: Evaluation on Safety of Self-titration in Insulin naïve People With Type 2 Diabetes Treated With Levemir® (Insulin Detemir) and Oral Antidiabetic Agents
Brief Title: Observational Study on Safety of Self-titration of Once Daily Levemir®
Acronym: SOLVE™
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3573
Record Dates: First submitted 2008-08-19; First posted 2008-08-25 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of a normal clinical evaluation.
  Other Names: NN304; Levemir®

SUMMARY:
This study is conducted in Europe. The main objective of the study is to assess the safety of self-titration in type 2 diabetic patients on antidiabetic tablets who are receiving insulin for the first time. The study will also look at the blood glucose control, frequency of dose adjustment, clinic visits, and time spent training patients to self-titrate.

The objective of diabetes management is to achieve blood glucose levels as close as possible to normal in order to avoid late stage diabetic complications. Self-titration (where patients adjust insulin dosage themselves) offers the potential for better blood glucose control than titration only at clinic visits. In recent years treatment of type 2 diabetes in the United Kingdom has moved from hospitals to GP surgeries or local clinics. Patients with type 2 diabetes, in general, have not been trained in self-titration to the same degree as patients with type 1 diabetes. Less experience in self-titration could impact the level of blood glucose control and outcome for these patients.

Data from this study will be pooled with data from NN304-3714 (NCT00825643) and will be reported in the final study report for NN304-3714.

ELIGIBILITY:
Inclusion Criteria:

* After the participating physician/nurse's decision has been made to initiate once daily Levemir® therapy (within the license of the product), any patient with type 2 diabetes of 18 years or older who is currently treated with diet, exercise and one or more OADs can be offered to participate

Exclusion Criteria:

* Patients unable to give written informed consent
* Current treatment with insulin
* Patient deemed unable or unwilling to self-titrate
* Known or suspected allergy to study product or related products
* Pregnancy or breastfeeding or intention of becoming pregnant within the next 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from a primary care setting who have been deemed appropriate to receive Levemir® as new treatment and as part of routine out-patient care by the prescribing health care professional.
Sampling Method: Non-Probability Sample
Enrollment: 882 (Actual)
Dates: Start 2008-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse drug reactions including major hypoglycaemic events | during treatment

SECONDARY OUTCOMES:
Incidence of serious adverse events and all adverse events | during treatment
Incidence of hypoglycaemic events | in the 4 weeks preceding the baseline, 12 and 20 week visits
HbA1c | at the interim study visit at 12 weeks and the end of the study visit at 20 weeks
Variability and mean of the patient's self-monitored plasma glucose measurements | at approximately 12 and 20 weeks
Proportion of patients who achieved equal or greater than 1% HbA1c reduction after initiation of insulin detemir without experiencing hypoglycaemic episodes | at approximately 12 and 20 weeks
Proportion of patients achieving FBG below 6.0 mmol/l +/- hypo | defined by the average of the last three FBGs
Body weight | at approximately 12 and 20 weeks
Frequency of insulin adjustment | at approximately 12 and 20 weeks
Total number of visits/contacts to the clinic, related to titration | at approximately 12 and 20 weeks
HCP time used on titration training | at baseline and approximately 12 and 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Crawley, United Kingdom

REFERENCES:
- [Result] Khunti K, Damci T, Meneghini L, Pan CY, Yale JF; SOLVE Study Group. Study of Once Daily Levemir (SOLVE): insights into the timing of insulin initiation in people with poorly controlled type 2 diabetes in routine clinical practice. Diabetes Obes Metab. 2012 Jul;14(7):654-61. doi: 10.1111/j.1463-1326.2012.01602.x. Epub 2012 Apr 22. PMID 22443213
- [Result] Ross S, Dzida G, Ji Q, Kaiser M, Ligthelm R, Meneghini L, Nazeri A, Orozco-Beltran D, Pan C, Svendsen AL; SOLVE Study Group. Safety of once-daily insulin detemir in patients with type 2 diabetes treated with oral hypoglycemic agents in routine clinical practice. J Diabetes. 2014 May;6(3):243-50. doi: 10.1111/1753-0407.12091. Epub 2013 Oct 29. PMID 24103141
- [Result] Vora J, Caputo S, Damci T, Orozco-Beltran D, Pan C, Svendsen AL, Solje KS, Khunti K; SOLVE study group. Effect of once-daily insulin detemir on oral antidiabetic drug (OAD) use in patients with type 2 diabetes. J Clin Pharm Ther. 2014 Apr;39(2):136-43. doi: 10.1111/jcpt.12116. Epub 2013 Dec 13. PMID 24329524
- [Result] Khunti K, Vora J, Davies M. Results from the UK cohort of SOLVE: providing insights into the timing of insulin initiation in people with poorly controlled type 2 diabetes in routine clinical practice. Prim Care Diabetes. 2014 Apr;8(1):57-63. doi: 10.1016/j.pcd.2013.11.010. Epub 2013 Dec 27. PMID 24378771
- [Derived] Khunti K, Damci T, Husemoen LL, Babu V, Liebl A. Exploring the characteristics of suboptimally controlled patients after 24weeks of basal insulin treatment: An individualized approach to intensification. Diabetes Res Clin Pract. 2017 Jan;123:209-217. doi: 10.1016/j.diabres.2016.11.028. Epub 2016 Dec 9. PMID 28061430
- [Derived] Orozco-Beltran D, Pan C, Svendsen AL, Faerch L, Caputo S; SOLVE Study Group. Basal insulin initiation in primary vs. specialist care: similar glycaemic control in two different patient populations. Int J Clin Pract. 2016 Mar;70(3):236-43. doi: 10.1111/ijcp.12776. Epub 2016 Feb 24. PMID 26916450
- [Derived] Damci T, Emral R, Svendsen AL, Balkir T, Vora J; SOLVE study group. Lower risk of hypoglycaemia and greater odds for weight loss with initiation of insulin detemir compared with insulin glargine in Turkish patients with type 2 diabetes mellitus: local results of a multinational observational study. BMC Endocr Disord. 2014 Jul 21;14:61. doi: 10.1186/1472-6823-14-61. PMID 25048824
- [Derived] Yale JF, Damci T, Kaiser M, Karnieli E, Khunti K, Liebl A, Baeres FM, Svendsen AL, Ross SA; SOLVE Study Group. Initiation of once daily insulin detemir is not associated with weight gain in patients with type 2 diabetes mellitus: results from an observational study. Diabetol Metab Syndr. 2013 Oct 2;5(1):56. doi: 10.1186/1758-5996-5-56. PMID 24499517
- [Derived] Liebl A, Andersen H, Svendsen AL, Vora J, Yale JF; SOLVE Study Group. Resource utilisation and quality of life following initiation of insulin detemir in patients with type 2 diabetes mellitus. Int J Clin Pract. 2013 Aug;67(8):740-9. doi: 10.1111/ijcp.12133. PMID 23869677
- [Derived] Karnieli E, Baeres FM, Dzida G, Ji Q, Ligthelm R, Ross S, Svendsen AL, Yale JF; SOLVE Study Group. Observational study of once-daily insulin detemir in people with type 2 diabetes aged 75 years or older: a sub-analysis of data from the Study of Once daily LeVEmir (SOLVE). Drugs Aging. 2013 Mar;30(3):167-75. doi: 10.1007/s40266-013-0054-3. PMID 23371395
- [Derived] Liebl A, Wilhelm B, Kaiser M. [Once daily insulin detemir in patients with type 2 diabetes: results of German centers in a 6-month international observational study (SOLVE)]. MMW Fortschr Med. 2012 Dec 17;154 Suppl 4:102-9. German. PMID 23326928
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com